CLINICAL TRIAL: NCT00570869
Title: Training Mothers of Infants in Infant Cardiopulmonary Resuscitation (CPR) Using a 22-Minute Instructional DVD and Infant Manikin
Brief Title: Training Mothers of Infants in Infant Cardiopulmonary Resuscitation (CPR)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lehigh Valley Hospital (Other)
Responsible Party: Principal Investigator, Marna Rayl Greenberg, Director of Emergency Medicine Research, Lehigh Valley Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2-20070911
Record Dates: First submitted 2007-12-10; First posted 2007-12-11 (Estimated); Last update posted 2012-04-26 (Estimated); Status verified 2012-04

CONDITIONS: Prevention of Sudden Death
Keywords: Infant CPR

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- CPR Class (Active Comparator): mothers who are currently certified in CPR (i.e., have taken the traditional CPR class, or have been recertified in CPR by classroom instruction, within the past two years).
  Interventions: Other: CPR Anytime

INTERVENTIONS:
Other: CPR Anytime — These participants will be consented, surveyed, asked to watch a 22-minute instructional Infant CPR DVD with an infant manikin.

SUMMARY:
This research will be a prospective, cohort study to determine if mothers of infants/newborns are more willing to complete CPR training using a 22-minute instructional DVD and infant manikin versus traditional four hour didactic instruction.

Study Hypothesis: A 22-minute instructional DVD and infant manikin will be an effective and preferred tool for teaching mothers of infants infant CPR.

Objectives

1. To determine if mothers of infants are more likely to complete infant CPR training with a 22-minute instructional DVD and infant manikin, than by attending a traditional CPR class.
2. To determine if learning infant CPR with a 22-minute instructional DVD and infant manikin is as effective as attending traditional infant CPR class.
3. To examine the number of mothers that were offered the opportunity to learn infant CPR either as part of their prenatal classes, or upon the birth of their infant.
4. To examine the number of mothers who have been previously trained in CPR.
5. To examine the reasons that mothers have been previously trained in CPR (e.g., mandated by work/career vs. personal reasons).
6. To examine the multiplier effect of an at home CPR education using a 22-minute instructional DVD and infant manikin at the time of the follow up phone call.

DETAILED DESCRIPTION:
This research will be a prospective, cohort study to determine if mothers of infants/newborns are more willing to complete CPR training using a 22-minute instructional DVD and infant manikin versus traditional four hour didactic instruction. Participants of the study will include mothers ages eighteen years and older, being treated as inpatients on the Mother Baby Unit (MBU) at the Cedar Crest (CC) site. Participants must have given birth within the last twenty-four hours, to a baby receiving care in the MBU nursery or the Neonatal Intensive Care Unit (NICU). Consent will be obtained from mother to participate. The control group will consist of those mothers who are currently certified in CPR (i.e., have taken the traditional CPR class, or have been recertified in CPR by classroom instruction, within the past two years). It is expected that this group will not have many participants because it is predicted that not many mothers will be certified in infant CPR prior to giving birth. After being consented, mothers will be surveyed, and tested on their CPR knowledge and proficiency before hospital discharge. The experimental group will consist of those participants who are not currently certified in CPR (i.e., have had traditional CPR training over two years ago which has lapsed, or who have never been certified in CPR). These participants will be consented, surveyed, asked to watch a 22-minute instructional DVD with an infant manikin, and then tested on CPR knowledge and proficiency before hospital discharge. Surveys will include questions pertaining to participant demographics, previous CPR learning experiences, reasons for obtaining and approximate cost of previous CPR instruction, and rating their instructional experiences (e.g., ease, quality of instruction, convenience, and effectiveness). Research staff will become CPR Instructors; and to ensure the inter-rater reliability each member of the staff will independently score CPR knowledge and performance in a series of mock CPR testing scenarios. During the study, research staff will be blinded to the group that the participants are enrolled in. Therefore, if one research staff member enrolls the participant, another blinded research staff member will assess the participants CPR proficiency in order to eliminate any instructor bias. Follow-up phone calls will be conducted 6 months post enrollment to measure the multiplier effect and to inquire about the incidence of having to use CPR skills in a real-life situation. Scores on participant's written and practical tests, responses to survey questions and follow up phone calls will be compared between groups.

ELIGIBILITY:
Inclusion Criteria:

1. Mother must be admitted to MBU at the CC site within twenty-four hours of giving birth.
2. Mother must be eighteen years-old or greater.

Exclusion Criteria:

1. Mother is not admitted to the MBU.
2. Mother is under eighteen years-old.
3. Mother has been inpatient for over twenty-four hours.
4. Mother is physically incapable of performing CPR.
5. Mother is cognitively impaired.
6. Mother is unable to understand and sign consent.
7. Mother is non-English speaking.
8. Current pregnancy resulted in fetal demise.
9. Mother who has previously participated in the study.
10. Mother who has previously self-educated themselves in infant CPR using a 22-minute DVD and an infant manikin.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2008-01; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Participants will be given written and practical exams to assess their learned CPR skills | 6 months

SECONDARY OUTCOMES:
CPR learning experiences (e.g., ease, quality of instruction, convenience, ) will be analyzed from survey results | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Marna R Greenberg, D.O., MPH, Principal Investigator — LVH
Locations (1):
- Lehigh Valley Hospital, Allentown, Pennsylvania, United States